CLINICAL TRIAL: NCT05040854
Title: Can we Rely on HLA to Predict Resistance to Biological Therapy in IBD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Hospitalar Tondela-Viseu (Other)
Responsible Party: Principal Investigator, Ana Carvalho, Principal Investigator, Centro Hospitalar Tondela-Viseu
Other Study IDs: CHTV07/2021.1
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Diseases; HLA; Biological therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples regarding inflammatory biomarkers and MHC class II
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Subjects: Blood donors
  Interventions: Genetic: HLA-DQA1*05 and DRB1
- IBD patients - under biological therapy: Patients with IBD followed up in consultation on biological therapy with anti-TNF, anti-integrin α₄β₇ or anti-interleukin 12-23.
  Interventions: Genetic: HLA-DQA1*05 and DRB1
- IBD patients - naive: Patients newly diagnosed with IBD and need for biological therapy with anti-TNF, anti-integrin α₄β₇ or anti-interleukin 12-23,
  Interventions: Genetic: HLA-DQA1*05 and DRB1

INTERVENTIONS:
Genetic: HLA-DQA1*05 and DRB1 — All patients will be asked to give blood samples to search for HLA-DQA1*05 and DRB1

SUMMARY:
The investigators propose an observational study including patients with inflammatory bowel disease under biological therapy with anti-TNF, anti-integrin α₄β₇ or anti-interleukin 12-23 (Ustekinumab), followed by an external Gastroenterology consultation at Centro Hospitalar Tondela-Viseu.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of IBD (according to ECCO diagnosis criteria);
* Adult patients (over 18 years);
* Full capability of signing informed consent.

Exclusion Criteria:

* Patients who refuse to participate in the study;
* Patients submitted to prior biological therapy (only for the IBD-naive group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Inflammatory Bowel Disease under biological therapy with anti-TNF, anti-integrin α₄β₇ or and anti-interleukin 12-23, followed in a gastroenterology outpatient consultation at the Centro Hospitalar Tondela-Viseu.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Response to biological therapy | 36 months
  To assess whether the presence of the HLA-DQA1*05 and HLA DRB1 alleles in patients with inflammatory bowel disease is associated with primary failure or loss of response to biological therapy with anti-TNF (Infliximab and Adalimumab), anti-integrin α₄β₇ (Vedolizumab) or anti-interleukin 12-23 (Ustekinumab).

SECONDARY OUTCOMES:
Prevalence of HLA-DQ1*05 and DRB1 | 36 months
  To determine the prevalence of HLA-DQ1*05 and DRB1 alleles in IBD population and to compare with a population of healthy blood donor patients.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Ministro, MD, Study Director — Centro Hospitalar Tondela-Viseu
Locations (1):
- Centro Hospitalar Tondela Viseu, Viseu, Portugal

REFERENCES:
- [Derived] Domingues A, Carvalho A, Martinho A, Soares C, Martins D, Sousa P, Araujo R, Cancela E, Silva A, Ministro P. Predicting resistance to biological therapy using human leukocyte antigen genes in patients with inflammatory bowel disease. Therap Adv Gastroenterol. 2025 Jul 11;18:17562848251353293. doi: 10.1177/17562848251353293. eCollection 2025. PMID 40655132